CLINICAL TRIAL: NCT05444582
Title: Levonorgestrel 52 mg IUD for Emergency Contraception and Same-Day Start
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00151440
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Contraception
Keywords: Emergency Contraception; IUD
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 52 mg LNG IUD Same Day Start or EC (Other): Week 1: Text daily for seven days. Report occurrences of the following in the last day: presence or absence of bleeding, spotting, pain, sexual intercourse, use of other methods of contraception, IUD expulsion or removal, and report any additional medical care received.
  Weeks 2 & 3: Weekly text survey assessing on which days of the previous week participants experienced bleeding and spotting, sexual intercourse, use of other methods of contraception, IUD expulsion or removal, or experienced adverse events.
  Week 4 Survey: At 28 days, participants will be asked about pregnancy symptoms, concern about pregnancy, and the result of their urine pregnancy test including a prompt to upload a photo of the test.
  Interventions: Drug: Levonorgestrel 52 MG Intrauterine System

INTERVENTIONS:
Drug: Levonorgestrel 52 MG Intrauterine System — Eligible participants must be 16-35 years old, meet clinic eligibility for IUD placement, and having a LNG 52 mg IUD placed for either:
  Emergency Contraception (had unprotected intercourse in the last 5 days) OR Same-day start - >7 days since the onset of last menstrual period and have no report of unprotected intercourse in the last 5 days.

SUMMARY:
This is a prospective clinical research study to test the effectiveness of the Levonorgestrel (LNG) 52 mg Intrauterine Device (IUD) for emergency contraception (EC) and same-day start use that will enroll people receiving care at Planned Parenthood affiliates across the U.S. Our prior work demonstrated efficacy (shows that it works in an ideal setting) for the LNG 52 mg IUD for these uses and this study will test effectiveness (how well it works in the real world) in a larger, heterogenous population in a usual care setting where participants select their method and are not randomly assigned to it. The study population will include people initiating an LNG 52 mg IUD and meet inclusion and exclusion criteria at 8 Planned Parenthood affiliates nationwide. Planned Parenthood Federation of America was the first major healthcare organization to change its practice to incorporate the changes we are studying here. As such, all study participants will be offered the opportunity to choose the interventional IUD at the site they visit. The primary outcome is pregnancy status one month after LNG IUD placement by home urine pregnancy test or clinical record review. Participant follow up concludes one month after enrollment.

The purpose of this study is to demonstrate reproducibility of earlier findings in a more heterogenous population. As such, IUD placement is not a study procedure but a component of clinical care. The study interventions only involve study participation and provision of data around the use of the levonorgestrel 52 mg IUD for EC or same day start.

DETAILED DESCRIPTION:
This protocol builds on our successful execution of the RAPID EC (RCT Assessing Pregnancy with Intrauterine Devices for Emergency Contraception) trial, which demonstrated the LNG 52 mg IUD to be noninferior to the copper IUD for EC. LNG 52 mg IUD users in the study had a one-month EC pregnancy rate of 0.3% (95% CI 0.01-1.7%). Within months of publication of these results in the New England Journal of Medicine, Planned Parenthood Federation of America's (PPFA) National Medical Committee used our data to adopt new contraceptive care guidelines. Today, those presenting for care at any of the over 600+ PPFA health centers in the U.S. can be provided the LNG 52 mg IUD for 2 new situations when they have a negative pregnancy test: 1) EC, within 5 days of unprotected intercourse (UPI) and; 2) Non-EC same-day start, at any point in the menstrual cycle without UPI in the last 5 days. PPFA's clinical application of these data removed an access barrier and will decrease people's risk of undesired pregnancy.

However, the LNG 52 mg IUD prescribing information and Centers for Disease Control and World Health Organization clinical guidelines, which guide clinical care outside of PPFA, currently oppose placement for both of these situations. The current recommendation for those not within the first 7 days of the menstrual cycle is to delay LNG IUD placement and return after the next menses start. We found in the RAPID EC trial and other analyses that the risk of pregnancy appears negligible when initiating an LNG 52 mg IUD for EC or same-day start, provided the urine pregnancy test is negative. This study assesses reproducibility of RAPID EC's findings by determining the effectiveness of the LNG 52 mg IUD to prevent pregnancy in real-world settings where users select their treatment (and are not randomized to it as in RAPID EC trial). We will test reproducibility and generalizability in a larger, more diverse population to assess the appropriateness of defining the interventional IUD as a new standard of care and how PPFA guidelines should be revised before influencing guidelines more broadly.

EC: Pills, the copper IUD, and the importance of adding the LNG 52 mg as a new EC option

Globally, people use EC methods to decrease their risk of pregnancy after UPI because of method failure or not using contraception. EC use in the U.S. is common and increasing. In 2002, 4% of pregnancy capable people ever reporting sexual intercourse had used EC. This figure climbed to 20% by 2015, and to 27% by 2017 for urban women. Although anyone can obtain oral EC without a prescription, IUDs can be desirable for EC because they are much more effective than EC pills and provide ongoing highly effective contraception for years if desired. So, while the majority of EC users do not want an IUD it is an important option with distinct benefits for those that do.

In the U.S., the Food and Drug Administration (FDA) has approved only two methods of EC: oral LNG and oral ulipristal acetate. A third method, the copper IUD, is an evidence-based EC approach and the most effective (failure rate <0.1%), with pregnancy risk an order of magnitude lower than the oral methods. However, those selecting an IUD for long-term contraception are more likely to choose the LNG over the copper IUD. Adding the LNG 52 mg IUD as another EC option, highly effective for both EC and ongoing contraception, is a significant advancement. Especially given that a greater number of contraceptive options presented to an individual is associated with increased method satisfaction, continuation, and decreased unintended pregnancy. The RAPID EC trial demonstrated efficacy for the first new EC method since the 2010 FDA approval of oral ulipristal acetate.

Oral EC methods are less effective in two critical situations where IUD EC efficacy does not change.

One, for people with a Body Mass Index (BMI) >30 kg/m2 the risk of pregnancy risk after oral EC rises to 2.6% for ulipristal users and to 5.8% for oral LNG EC users, approaching no effect. However, IUD pregnancy risk does not change with weight for either EC (half of RAPID EC participants had a BMI 25 or greater) or ongoing contraception. Public health significance of this issue increases as the mean BMI for U.S. women of reproductive age rises toward 30 kg/m2. Two, the absolute highest risk of pregnancy for oral LNG EC users, 7.3%, is in women reporting additional acts of intercourse later in the cycle after EC use. This elevated risk of pregnancy is eliminated when an IUD is placed for EC as supported by a RAPID EC secondary analysis.

Same-day LNG IUD start reduces ongoing pregnancy risk and promotes autonomy.

"Same-day start" describes the need to provide people their desired method of contraception on the day they present for care. Meeting people's needs on the day they present for care is important because requiring two visits for IUD placement for STI testing, which is unnecessary to reduce infection risk, or additional counseling sessions, results in only half (54%) returning to get the IUD. Adolescents, post-abortion, and postpartum patients who receive long acting reversible contraceptive (LARC) methods when presenting for care, rather than returning later, are more likely to get their desired method and have lower pregnancy rates. Same-day LARC access is supported by The American College of Obstetricians and Gynecologists, but is only provided by 29% of U.S. Obstetrician Gynecologists.

Provision of the LNG IUD for EC and same-day start use is an important step in removing access barriers to contraception and providing people with the method they desire at the time that they present for care. We hypothesize both reproducibility of the initial results and greater generalizability. This effectiveness study will expand on the previous trial, conducted in one geographic area, by enrolling a heterogeneous participant population from 8 U.S. PPFA affiliates, providing geographic, racial, ethnic, and gender diversity.

ELIGIBILITY:
Inclusion Criteria:

* Meet clinic eligibility for IUD placement
* Have a LNG 52 mg IUD placed for either emergency contraception (had unprotected intercourse in the last 5 days) OR Same-day start, >7 days since the onset of last menstrual period and have no report of unprotected intercourse in the last 5 days
* Negative high sensitivity urine pregnancy test prior to IUD placement.
* No known contraindications to the LNG 52 mg IUD per the CDC Medical Eligibility Criteria for Contraceptive Use 2016
* Have had penile-vaginal intercourse at least once since their last menstrual period. If last menstrual period is unknown or irregular, then have had penile-vaginal intercourse at least once in the last month.
* Fluent in English or Spanish
* Working Cell Phone number that receives text messages
* Willing to comply with the study requirements including providing 1-month follow up data including a urine pregnancy test result one month after IUD placement

Exclusion Criteria:

* Current pregnancy
* Currently Breastfeeding
* Current use of permanent contraception (has had a hysterectomy, tubal permanent contraception, or partner with a vasectomy in the last month)
* Use of any contraceptive pills, patches, vaginal rings or any contraceptive implant or IUD use in the last 4 weeks
* Use of oral emergency contraception in last 5 days
* Vaginal bleeding of unknown etiology
* Use of injectable hormonal contraceptive (Depo-Provera) in the last 6 months
* Planned use of any non-contraceptive estrogen, progesterone, or testosterone
* Acute cervicitis
* Known abnormalities of the uterus that distort the uterine cavity
* Ended pregnancy at or under 20 weeks gestational age within the last 2 weeks
* Ended pregnancy over 20 weeks gestational age within the last 6 weeks

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1404 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of pregnancies reported in participants at one month post insertion of IUD | One Month
  Positive pregnancies reported by participants through survey and photo of pregnancy test one month after LNG IUD placement by home urine pregnancy test or clinical record review.

SECONDARY OUTCOMES:
Percentage of participants continuing to use IUD at one month post insertion | One Month
  Percentage of participants continuing to use IUD at one month post insertion

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, MPH, Principal Investigator — University of Utah
Locations (8):
- United States (8):
  - Planned Parenthood Mar Monte, San Jose, California
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Planned Parenthood Illinoi, Chicago, Illinois
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Planned Parenthood North Central States, Saint Paul, Minnesota
  - Planned Parenthood Columbia Willamette, Portland, Oregon
  - Planned Parenthood Association of Utah, Salt Lake City, Utah
  - Planned Parenthood Great Northwest Hawaii, Alaska, Indiana, Kentucky, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No